CLINICAL TRIAL: NCT00392132
Title: Impact of Screening Patients With HIV for Kidney Disease
Status: Withdrawn | Type: Observational
Why Stopped: Sufficient study funding was not obtained.
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Darren Schmidt, Assistant Professor of Medicine, University of Mississippi Medical Center
Other Study IDs: UMMC - HIV and CKD
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: HIV Infections; Renal Insufficiency, Chronic; Proteinuria
Keywords: HIV
MeSH Terms: conditions — HIV Infections; Renal Insufficiency, Chronic; Proteinuria

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The Infectious Disease Society of America has recently recommended that patients with Human Immunodeficiency Virus (HIV) be screened for kidney disease on a regular basis. Screening involves non-invasive urine and blood test and a screening program has already been initiated here in the University of Mississippi HIV clinic. This study looks at the effect of this new screening program. Our Hypothesis is that screening for kidney disease is a cost effective and important addition to the care of patients with HIV.

DETAILED DESCRIPTION:
The Infectious Disease Society of America has recently recommended that patients with Human Immunodeficiency Virus (HIV) be screened for kidney disease on a regular basis. Screening involves non-invasive urine and blood test and a screening program has already been initiated here in the University of Mississippi HIV clinic. However nobody knows for sure whether this will help doctors take better care of patient with HIV.

This study looks at the effect of this new screening program. We want to see how frequently abnormalities are seen on screening, how frequently certain kidney diseases are diagnosed, how often patients are referred to a nephrologist and how often a patient's management is changed by the screening. We will also estimate the cost-benefit ratio of the screening. We will review patient charts to determine what has happened in each case where screening was conducted.

This study will not involve any additional testing.

The benefit of this study will be improving our understanding of kidney disease in HIV. It will help us determine the value of screening for kidney disease and the frequency of certain kidney diseases in HIV in our clinic population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with HIV who are seen by the University of Mississippi Infectious disease clinic at the Jackson Medical Mall or patient seen at the University of Mississippi Nephrology Clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Primary Completion 2006-10 (Estimated); Study Completion 2006-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Darren W Schmidt, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States